CLINICAL TRIAL: NCT02863900
Title: From the Characterization of the Cholesterol-epoxide Pathway Deregulation to New Therapeutic Perspectives in Breast Cancers
Acronym: BREASTEROL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 16SEIN04
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental arm (Experimental): subtypes of BC (namely luminal A and luminal B, HER2+, TN)
  Interventions: Other: cohort of BC of each subtypes

INTERVENTIONS:
Other: cohort of BC of each subtypes

SUMMARY:
The main objective of our project is to further characterize the deregulation of CE (Cholesterol Epoxides) metabolism in different moleculars subtypes of BC (BC=Breast Cancer) (luminal A and B, HER2+ and triple negative). We will study not only the level of expression of the enzymes involved in this pathway by immuno-histochemistry, all the enzymes involved were identified in our preclinical work (GSTA1 (Glutathione S-Transferase A1 ), DHCR7, D8D7I, 11βHSD2 (11β-hydroxysteroid dehydrogenase of type 2 )), but also the metabolite rates of CE (hydrolyses cholesterols-5,6-epoxide ), CT (into cholestane-3β, 5α, 6β triol ), DDA (Dendrogenin A)and OCDO (6-oxo-cholestan-3β, 5α-diol ). Our preliminary results demonstrate the feasibility of these dosages. We will also establish whether these deregulations are i) correlated with different histo-prognostic parameters (pN (N= Node), pT (T= Tumor) , EV, TIL…) but also clinical ii) an independent prognostic parameter of BC in terms of disease-free survival, metastasis-free survival and overall survival. The cohort consists of 350 cases of BC, treated between 2009 and 2011 as well as all relevant clinical informations. In parallel, we will continue our preclinical work by characterizing the targets and mechanisms of action of OCDO. Our preliminary results indicate that OCDO is a modulator of the glucocorticoid receptor (GR), which could be target to inhibit this pathway. On the other hand, we will characterize in the same manner as in human tumors, the deregulations of the CE metabolism in vitro and in vivo (including xenografts in mice of human tumors, in collaboration with Roman-Roman S) on a representative panel of BC molecular subtypes, sensitive or not usually administered in clinical treatment and study the anti-tumor effect of various "anti-OCDO" therapies (therapies preventing its production such as Tam (tamoxifen) or DDA, inhibitor of the enzyme producing OCDO, or an inhibitor of the GR (glucocorticoid receptor )), alone or in combination with conventional therapies

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Affiliated to the French social security system.
* Subjects must provide written informed consent prior to any study-specific procedure or assessment

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Subject law protected
* Any serious and/or unstable pre-existing psychiatric,familial, geographic or social condition that could interfere with medical follow-up and compliance to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of the deregulations of CE metabolism in the different molecular subtypes of BC (namely luminal A and luminal B, HER2+, TN) | up to 3 years

SECONDARY OUTCOMES:
Compare CE metabolism characterisation and immune infiltrate by quantification of TILs (infiltrating-lymphocytes) | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Florence DALENC, MD, Principal Investigator — Institut Claudius Regaud
Locations (1):
- Institut Claudius Regaud, Toulouse, France

IPD SHARING:
Plan to Share IPD: No